CLINICAL TRIAL: NCT06247800
Title: Virtual Reality: Satisfaction and Tolerability as a Distraction During Small Bore Intercostal Chest Drain Insertion an Open Label Randomized Control Trial
Brief Title: Virtual Reality: Distraction During Small Bore Intercostal Chest Drain Insertion
Acronym: VR-STICH
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: National University of Malaysia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: FF-2024-002
Record Dates: First submitted 2024-01-15; First posted 2024-02-08 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Pleural Effusion
MeSH Terms: conditions — Pleural Effusion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patient undergoing chest drain with the use of VR device (Active Comparator): Patient undergoing chest drain with the use of VR device on, for those on VR device, they will be shown a video consisting of calming nature scene together with soothing instrumental music.
  Interventions: Device: Virtual Reality Device
- Patient undergoing chest drain without the use of VR device (Active Comparator): Patient undergoing chest drain without the use of VR device on, as per standard practise
  Interventions: Other: Without virtual reality

INTERVENTIONS:
Device: Virtual Reality Device — A virtual reality headset is a heads-up display that allows users to interact with simulated environment.
  Arms: Patient undergoing chest drain with the use of VR device
Other: Without virtual reality — Patients undergoing intercostal chest drain without the use VR device
  Arms: Patient undergoing chest drain without the use of VR device

SUMMARY:
Intercostal chest drain (ICC) insertion is a common procedure done worldwide to treat and diagnose pleural disease. It is used to evacuate fluid, blood, or air in the cavity from a myriad of causes namely pleural effusions of different etiologies, empyema, hemothorax, chylothorax and pneumothorax. It also functions as a route for antibiotics, pleurodesis and fibrinolytics. Hippocrates, whose practiced medicine 2,400 years ago, is often credited with being the first to insert a metal tube into the pleural region to drain fluid. It wasn't until the 19th century that a closed drainage system was properly documented in the literature, although open drainage remained to be the norm for quite some time.

In the past, large-bore tubes (24-32 F) were recommended in nearly all circumstances and were inserted using a blunt dissection technique. However, during the past two decades, small-bore catheters have become increasingly popular. They were first used to drain abdominal collections and have now been adopted for use in draining the pleural cavity utilizing the needle and guide wire Seldinger procedure, typically with radiological guidance. In addition to that, Seldinger technique allow us to insert the catheter at lower intercostals spaces without injury to the diaphragm or abdominal organs, thereby ensuring patient safety.

DETAILED DESCRIPTION:
Research Questions Can Virtual Reality serve as a diversion and improve participant's satisfaction and tolerability during the insertion of a small-bore intercostal chest drain?

Hypothesis VR leads to better satisfaction of participant during ICC insertion VR reduce pain and anxiety during ICC insertion VR leads to better satisfaction of proceduralist during ICC insertion

Type of Study This is a single center, prospective, interventional study of in-patient participants who are diagnosed with pleural disease and under follow up Respiratory Unit Hospital Canselor Tuanku Muhriz, Universiti Kebangsaan Malaysia. All participants involved in the study will be randomized by 4 block randomizations into either interventional group (VR) or control group (without VR). All participants will be undergoing small bore ICC drain on top of standard care during procedure.

Demographic data was collected prior to randomization, which included (age, gender, ethnicity, BMI, comorbidities) and indications for ICC. The investigator then randomized into 2 groups via block randomization into intervention (VR) and controlled group (without VR).

Subsequently, consent will be obtained from those who are agree to participate, either from the participant him/herself or their next-of-kin. The process of briefing and obtaining consent will be only done once the participant is stable. These processes will not in any way interfering with clinical evaluation, investigation, treatment and intervention done to the participant by the attending doctor. All of the consented participants will be undergoing ICC insertion.

Prior to the ICC insertion, vital signs will be recorded and both groups will be given a VAS questionnaire to assess their pain and breathlessness. This is done to determine the participant's baseline score pre-procedure. The pain score was measured by the use of validated 10 cm VAS, a 10 cm line anchored with "no pain" at 0 cm and "unbearable pain" at 10 cm. The breathlessness VAS was measured with a similar scale which was anchored with "no breathlessness" at 0 cm, and "worst possible breathlessness" at 10 cm. Participants will also be given State-Trait-Anxiety-Inventory (STAI) questionnaire. It comprised of twenty statements that assess how respondents feel "at the present time.". They were instructed to circle the number that describes the intensity of their feelings concerning each question best: 1, "not at all;" 2, "somewhat;" 3, "moderately so;" 4, "very much so.". The STAI has a potential score range spanning from 20 to 80, and our study employed both English and a verified translated version in Malay for the questionnaire.

After completing the questionnaires, participants in the interventional group will be given the virtual reality (VR) device to wear, which was the Oculus Quest 2 (Oculus, China) before ICC insertion. The device is owned by respiratory unit HCTM and had been utilized in previous study. Videos of natural scenery were played for them while calming instrumental music played in the background. Three-dimensional footage of natural landscapes from across the world was played as participants listened to instrumental music through surround sound speakers. The participants were given ten minutes of screening time prior to performing ICC, and after ICC insertion was complete, the device was withdrawn. The VR device was sanitized before and after each use, and participants were given disposable hygiene covers to prevent the risk of pathogen transmission.

Local anaesthesia will be given as to the participants prior to the procedure at the site of insertion. ICC insertion will be performed by 2 proceduralist with a 3-year experience in performing ICC. Post-procedure, VAS questionnaires will be given to participant (on pain and breathlessness), STAI questionnaire on anxiety and satisfaction questionnaire (Likert's scale). These will be completed by the participants at 30 min post procedure. Vital signs of participant will also be taken and recorded post procedure. The proceduralist will be given satisfaction questionnaire upon completion of procedure

ELIGIBILITY:
Inclusion Criteria:

* All participants undergoing ICC insertion
* Participants who could understand and give consent

Exclusion Criteria

* Participants who are unable to understand or give consent
* Ventilated patients
* Participants who are not comfortable wearing VR device
* Participants who are unable to communicate (illiterate, had hearing impairment, mute, blind or had memory impairment)
* Participants with craniofacial deformity
* Participants who are on sedative medication

Traumatic or post Motor Vehicular Accident patient Participants undergoing Indwelling pleural catheter insertion Participants with anxiety disorder

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2026-12-25 (Estimated); Study Completion 2026-12-25 (Estimated)

PRIMARY OUTCOMES:
To compare the satisfaction of participants undergoing intercostal chest drain insertion with or without VR using a 5-point Likert scale satisfaction questionnaire (1 - very dissatisfied, 2-dissatisfied, 3-neutral, 4-satisfied, 5-very satisfied). | 30 minutes after procedure
  Participants who underwent intercostal chest drain insertion with and without VR device will be assess with 5 point Likert Scale for satisfaction score.

SECONDARY OUTCOMES:
To assess tolerability (pain, and breathlessness) of participants undergoing ICC with or without VR, using a 10 cm Visual analogue scale (VAS), ranging from 0 (no bother) to 10 (worst intolerable level) before ICC insertion | 10 minutes before procedure
  Participants undergoing intercostal chest drain insertion with and without VR device will be assessed with VAS Score to assess tolerability
To assess tolerability (pain, and breathlessness) of participants undergoing ICC with or without VR, using a 10 cm Visual analogue scale (VAS), ranging from 0 (no bother) to 10 (worst intolerable level) after ICC insertion | 30 minutes after procedure
  Participants undergoing intercostal chest drain insertion with and without VR device will be assessed with VAS Score to assess tolerability
To assess the anxiety of participants undergoing ICC with or without VR using the State-Trait-Anxiety-Inventory (STAI) score before ICC insertion (minimum score of 20 to maximum score of 80) | 10 minutes before procedure
  Participants undergoing intercostal chest drain insertion with and without VR device will be assessed with STAI Score to assess anxiety
To assess the anxiety of participants undergoing ICC with or without VR using the State-Trait-Anxiety-Inventory (STAI) score after ICC insertion (minimum score of 20 to maximum score of 80) | 30 minutes before procedure
  Participants undergoing intercostal chest drain insertion with and without VR device will be assessed with STAI Score to assess anxiety
To assess satisfaction of proceduralist's performing ICC insertion with or without VR using satisfaction questionnaire (5-point Likert scale). (1 - very dissatisfied, 2-dissatisfied, 3-neutral, 4-satisfied, 5-very satisfied). | 30 minutes after procedure
  Procedurist will be given 5-point Likert Scale to assess satisfaction in performing intercostal chest drain device
To assess Systolic and Diastolic Blood pressure (in mmHg) , of participants undergoing ICC with and without VR at before ICC insertion | 5 minute before procedure
  Participants' vital sign will be assessed at baseline before ICC insertion
To assess Systolic and Diastolic Blood pressure (in mmHg) , of participants undergoing ICC insertion with and without VR after ICC insertion | 5 minute after procedure
  Participants' vital sign will be assessed after ICC insertion
To assess Heart rate (rates/minute) of participants undergoing ICC insertion with and without VR at before ICC insertion | 5 minute before procedure
  Participants' vital sign will be assessed at baseline before ICC insertion
To assess Heart rate (rates/minute) of participants undergoing ICC insertion with and without VR after ICC insertion | 5 minute after procedure
  Participants' vital sign will be assessed after ICC insertion

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Faisal Abdul Hamid, MBBS (IIUM), Principal Investigator — National University of Malaysia
Locations (1):
- National University of Malaysia, Kuala Lumpur, Kuala Lumpur, Malaysia

IPD SHARING:
Plan to Share IPD: No